CLINICAL TRIAL: NCT05811403
Title: The Influence of Epigallocatechin Gallate (EGCG) as a Flushing Agent During Full Pulpotomy Using Two Different Calcium Silicate-based Materials on Postoperative Pain and Success Rate in Mature Permanent Molars With Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Epigallocatechin Gallate (EGCG) as a Flushing Agent During Full Pulpotomy in Mature Permanent Molars With Irreversible Pulpitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Anan Medhat Mohamed, Assistant lecturer, Ahram Canadian university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 372
Record Dates: First submitted 2023-03-18; First posted 2023-04-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Irreversible Pulpitis
MeSH Terms: interventions — epigallocatechin gallate; Sodium Hypochlorite; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator will not be blinded because of the nature of the intervention and comparator (the flushing agent and pulp capping material)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EGCG as a flushing fluid, MTA as a pulp capping material (Experimental)
  Interventions: Other: Epigallocatechin gallate (EGCG); Other: Mineral trioxide aggregate (MTA)
- EGCG as a flushing fluid, Premixed BC putty as a pulp capping material (Experimental)
  Interventions: Other: Epigallocatechin gallate (EGCG); Other: Premixed bioceramic putty
- NaOCl as a flushing fluid, Premixed BC putty as a pulp capping material (Experimental)
  Interventions: Other: Sodium hypochlorite (NaOCl); Other: Premixed bioceramic putty
- NaOCl as a flushing fluid, MTA as a pulp capping material (Active Comparator)
  Interventions: Other: Sodium hypochlorite (NaOCl); Other: Mineral trioxide aggregate (MTA)

INTERVENTIONS:
Other: Epigallocatechin gallate (EGCG) — Epigallocatechin gallate (EGCG) is a white powder that can be obtained from tea leaves. It accounts for 50-60 % of catechin content of tea polyphenols with a wide range of biological activities including antioxidant, antimicrobial, anti-inflammatory, immune regulatory, anti-tumour effects.
  Arms: EGCG as a flushing fluid, MTA as a pulp capping material; EGCG as a flushing fluid, Premixed BC putty as a pulp capping material
Other: Sodium hypochlorite (NaOCl) — Sodium hypochlorite (NaOCl) is an excellent non-specific proteolytic and antimicrobial agent that provides disinfection of the dentin-pulp interface.
  Arms: NaOCl as a flushing fluid, MTA as a pulp capping material; NaOCl as a flushing fluid, Premixed BC putty as a pulp capping material
Other: Mineral trioxide aggregate (MTA) — Mineral trioxide aggregate (MTA) is the material of choice for pulp capping in vital pulp therapy.
  Arms: EGCG as a flushing fluid, MTA as a pulp capping material; NaOCl as a flushing fluid, MTA as a pulp capping material
Other: Premixed bioceramic putty — Bioceramic putty is a premixed, ready-to-use calcium silicate-based material which can be used as a pulp capping material.
  Arms: EGCG as a flushing fluid, Premixed BC putty as a pulp capping material; NaOCl as a flushing fluid, Premixed BC putty as a pulp capping material

SUMMARY:
This study evaluates the effect of two flushing agents (epigallocatechin gallate (EGCG) and sodium hypochlorite (NaOCl)) during full pulpotomy using two different calcium silicate-based materials (MTA and premixed bioceramic putty) on postoperative pain, success rate and dentin bridge thickness in mature permanent mandibular molars with irreversible pulpitis. Participants will be divided into four groups based on the flushing fluid and the pulp capping material to be used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either gender between the age group of 20-40 years.
2. Systemically healthy patient (ASA I or II).
3. Mature permanent mandibular molars with:

   * Extremely deep carious lesion (caries penetrating entire thickness of dentin).
   * Clinical diagnosis of symptomatic irreversible pulpitis and normal periapical tissue.
4. Patients who agree to provide written consent and attend for recall appointments.

Exclusion Criteria:

1. Non-restorable teeth with subgingival caries or badly broken teeth.
2. Signs of pulpal necrosis; associated sinus tract or swelling.
3. Negative response to pulp sensibility test.
4. Poor periodontal support.
5. Absence of pulp exposure following complete caries removal.
6. Bleeding from the pulp could not be detected from one or more of the orifices indicating pulp necrosis.
7. Failure to achieve haemostasis within 10 min following full pulpotomy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | One week
  Pain assessments will be made at 24, 48, 72 hours and one week postoperatively using an 11-point NRS. Pain will be categorized into 4 categories as follows: 0 reading represents "no pain"; 1- 3 readings represent "mild pain"; 4- 6 readings represent "moderate pain"; 7- 10 readings represent "severe pain".

SECONDARY OUTCOMES:
Clinical success | One year follow-up
  The outcome will be considered successful in case of absence of clinical signs and symptoms indicative of pulpal or periapical pathosis (pain and tenderness to percussion).
Radiographic success | One year follow-up
  The outcome will be considered successful in case of complete radiographic healing (PAI score 1 or 2) with absence of any pathosis on recall radiographs such as root resorption.
Dentin bridge thickness | 12 months
  CBCT scans will be performed at 12 months to measure the thickness of the dentin bridge formed at the interface between the pulp capping material and the radicular pulp.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided